CLINICAL TRIAL: NCT04143958
Title: A Randomized, Open-label, Active Comparator, 2-arm, Prospective Study to Assess the Glycosphingolipid Clearance and Clinical Effects of Switching to Agalsidase Beta (Fabrazyme) Versus Continuing on Agalsidase Alfa (Replagal) in Male Patients With Classic Fabry Disease
Brief Title: To Assess the Glycosphingolipid Clearance and Clinical Effects of Switching to Agalsidase Beta (Fabrazyme) Versus Continuing on Agalsidase Alfa (Replagal) in Male Patients With Classic Fabry Disease
Acronym: BCLEAR1
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The Sponsor terminated the study due to recruitment infeasibility without having enrolled any patient.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS15918; 2019-000064-21 (EudraCT Number); U1111-1223-5105 (Other: UTN)
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase beta; agalsidase alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- agalsidase beta (Experimental): Commercially available agalsidase beta treatment at approved dose and regimen;administered once every 2 weeks as an IV infusion
  Interventions: Drug: agalsidase beta (GZ419828)
- agalsidase alfa (Active Comparator): Commercially available agalsidase alfa treatment at approved dose and regimen; administered once every 2 weeks as an IV infusion
  Interventions: Drug: agalsidase alfa

INTERVENTIONS:
Drug: agalsidase beta (GZ419828) — Pharmaceutical form:Powder for concentrate for solution for infusion Route of administration: Intravenous (IV) infusion,
  Arms: agalsidase beta
Drug: agalsidase alfa — Pharmaceutical form:concentrate for solution for infusion Route of administration: Intravenous (IV) infusion
  Arms: agalsidase alfa

SUMMARY:
Primary Objective:

To assess reduction of plasma lyso-GL3 level after switch to agalsidase beta from agalsidase alfa

Secondary Objectives:

* To assess reduction of kidney podocyte GL3 content after switch to agalsidase beta from agalsidase alfa
* To assess reduction of GL3 content in endothelial skin cells after switch to agalsidase beta from agalsidase alfa
* To assess change in renal function after switch to agalsidase beta from agalsidase alfa
* To assess disease severity and clinical changes after switch to agalsidase beta from agalsidase alfa
* To assess improvement in symptoms of Fabry disease after switch to agalsidase beta from agalsidase alfa

DETAILED DESCRIPTION:
The study will have a screening period of up to 9 weeks. Eligible participants will be randomized to switch to agalsidase beta or to continue agalsidase alfa in a 1:1 ratio for a period of 12 months (52 weeks).

ELIGIBILITY:
Inclusion criteria :

* Male participant must be 16 to 45 years of age inclusive, at the time of signing the informed consent.
* Participants who are diagnosed with classic Fabry disease based on phenotype, presence or absence of characteristic Fabry disease symptoms including neuropathic pain, clustered angiokeratoma and/or cornea verticillata, leucocyte α-GAL A enzyme activity (3% or less compared to control), and genotype (optional).
* Participants who are currently receiving agalsidase alfa for a minimum of 6 months at an average dose of 0.2 mg/kg every other week (ie, every 2 weeks) at baseline.
* Participants who are naïve to agalsidase beta.
* Participants with estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73 m^2 at screening and baseline.
* Proteinuria level as measured by 2 separate, morning, clean-catch urine samples taken a few days apart demonstrating an averaged urine protein-creatinine ratio of <0.5 (ie, <500 mg protein per 1 g creatinine) between the 2 samples. For participants on angiotensin-converting enzyme inhibitors (ACEIs) or angiotensin receptor blockers (ARBs), the criterion is to be met both prior and after a temporary interruption of ACEIs/ARBs for 4 weeks.
* Participants with plasma lyso-GL3 levels >20 ng/mL on 2 consecutive samples taken at least 4 weeks apart.
* Participant's medical records (including eGFR values) available and accessible during the study period.
* Participant and/or participant's legal representative has given signed informed consent as described in the protocol which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. For potential participants age 16 to 18 years, a parent or legal representative is required to sign the ICF, and the potential participant is also required to sign an informed assent form.

Exclusion criteria:

* Participants with severe renal impairment (end-stage renal disease, dialysis, or renal transplantation) and/or nephropathies (including diabetic).
* Participants with rapid renal decline: Loss of >6mL/min/1.73 m^2 at screening compared to the most recent eGFR value approximately 12 months prior to screening.
* Participants with advanced cardiac failure (Stage D).
* Participants with bleeding disorder, prior history of unexplained bleeding episodes, or receiving mandatory anticoagulants or antiplatelets for any indication not allowing interruption of therapy for renal biopsy.
* Participants with diagnosed diabetes.
* Participants with history of anaphylaxis to Enzyme Replacement Therapy (ERT).
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study.
* Participants treated for more than 5 years with agalsidase alfa at an average dose of 0.2 mg/kg every other week (ie, every 2 weeks) prior to randomization.
* Exposure to migalastat or any investigational study intervention, except agalsidase alfa, for Fabry disease in the last 5 years prior to study participation. Patients who previously participated in any agalsidase alfa clinical study will be eligible if they meet other criteria.
* Exposure to any investigational drugs in the last 4 weeks or 5 half-lives, whichever is longer, prior to screening visit or concomitant enrollment in any other clinical study involving an investigational study treatment.
* Individuals accommodated in an institution because of regulatory or legal order; prisoners or subjects who are legally institutionalized.
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures.
* Participants are dependent on the Sponsor or Investigator or deemed vulnerable for any reason (in conjunction with Section 1.61 of the International Council for Harmonisation Good Clinical Practice [ICH-GCP] Ordinance E6).
* Participants who are employees of the clinical study center or other individuals directly involved in the conduct of the study, or immediate family members of such individuals.
* Any specific situation during study implementation/course that may raise ethics consideration

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 16 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Change in Plasma globotriaosylsphingosine (lyso-GL3) level | Baseline, 12 months (week 52)
  Change from baseline to 12 months (week 52) for plasma lyso-GL3 level

SECONDARY OUTCOMES:
Change in GL3 content in podocytes | Baseline, 12 months (week 52)
  Change from baseline to 12 months (week 52) for GL3 content in podocytes
Change in GL3 content in endothelial skin cells | Baseline, 12 months (week 52)
  Change from baseline to 12 months (Week 52) for GL3 content in endothelial skin cells
Change in measured glomerular filtration rate (mGFR) | Baseline, 12 months (week 52)
  Change from baseline to 12 months (Week 52) for measured glomerular filtration rate (mGFR) (measured by iohexol clearance)
Change in estimated glomerular filtration rate (eGFR) calculated | Baseline, 12 months (week 52)
  Change from baseline to 12 months (Week 52) for estimated glomerular filtration rate (eGFR) calculated using age appropriate formula [Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)/ Bedside-Schwartz]
Change in Mainz Severity Score Index (MSSI) total score | Baseline, 12 months (week 52)
  Change from baseline to 12 months (Week 52) for Mainz Severity Score Index (MSSI), based on MSSI total score
Change in Fabry Disease Patient Reported Outcomes (FD-PRO) total symptom score | Baseline, 12 months (week 52)
  Change from baseline to 12 months (Week 52) in Fabry Disease Patient Reported Outcomes (FD-PRO) score, based on FD-PRO total symptom score

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org